CLINICAL TRIAL: NCT02158169
Title: Pharmaco-epidemiological Study on the Effect of Retacrit® on Chemotherapy Induced Anaemia in Standard Oncology and Haematology Practice: Impact of Concomitant Iron Supplementation
Brief Title: Biosimilar Retacrit® in the Treatment of Chemotherapy-induced Anaemia in Oncology and Haematology
Acronym: SYNERGY
Status: Completed | Type: Observational
Sponsor: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: Synergy
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Chemotherapy-induced Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to describe, in a real-life context, the impact of an epoetin alpha biosimilar, Retacrit®, on anaemia in patients receiving chemotherapy, according to concomitant iron supplementation.

DETAILED DESCRIPTION:
This is a longitudinal, observational, prospective, multicentre, cohort study, conducted on a representative sample of public and/or private hospital-based oncologists and haematologists practicing in Metropolitan France.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, aged 18 years and older, seen by the oncologist or hematologist for chemotherapy.
* Patients for whom the oncologist or hematologist has decided the initiation of an epoetin alpha biosimilar treatment (Retacrit®) for anemia.
* Patients informed about the computer processing of their medical data and their right of access and correction.

Exclusion Criteria:

* Patients with hemoglobin concentrations >11 g/dL.
* Patients who have been transfused within the previous month.
* Patients who are hypersensitive to erythropoietin or one of its excipients.
* Patients participating or having participated in the previous month in a clinical trial in the field of anaemia in oncology.
* Patients refusing to participate in the observational study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients for whom the oncologist decides to initiate epoetin alpha biosimilar treatment (curative or prophylactic) will be asked to participate from treatment initiation (baseline visit) up to 12-16 weeks after inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 2167 (Actual)
Dates: Start 2012-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Impact of an epoetin alpha biosimilar with or without iron supplementation on chemotherapy-induced anemia | Patients are included at the time of the epoetin alpha biosimilar treatment initiation for chemotherapy-induced anemia and followed up to 12 to 16 weeks
  The efficiency of epoetin alpha biosimilar will be assessed by the responders'rate according to European Society for Medical Oncology (ESMO) guidelines. This rate will be compared depending on the iron supplementation.
  The safety will be assessed by the record of adverse effects (serious or not) and treatment discontinuation.

SECONDARY OUTCOMES:
Characteristics of patients receiving treatment with an epoetin alpha biosimilar, Retacrit®, for chemotherapy induced anaemia | Baseline visit
Procedures for evaluating possible iron deficiency and iron supplementation | At 12 to 16 weeks from baseline or at the end of chemotherapy
Impact of iron supplementation on the doses of Retacrit® used, and on treatment duration | At 12 to 16 weeks from baseline or at the end of chemotherapy
Experience of patients treated with Retacrit® | At 12 to 16 weeks from baseline or at the end of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Hélène ALBRAND, MD, Study Director — Hospira, now a wholly owned subsidiary of Pfizer
Locations (69):
- France (69):
  - Hopital Louis Pasteur, Colmar, Alsace
  - CH Emile Muller, Mulhouse, Alsace
  - CAC Paul Strauss, Strasbourg, Alsace
  - Chu Hopital Civil, Strasbourg, Alsace
  - MEDIPOLE, Aix-les-Bains, Auvergne-Rhône-Alpes
  - CHRA, Annecy, Auvergne-Rhône-Alpes
  - Clinique CONVERT, Bourg-en-Bresse, Auvergne-Rhône-Alpes
  - Ch Chambery, Chambéry, Auvergne-Rhône-Alpes
  - Chu Grenoble, Grenoble, Auvergne-Rhône-Alpes
  - Ch Valence, Valence, Auvergne-Rhône-Alpes
  - Chu Rennes, Rennes, Basse Normandie
  - CHU SUD, Rennes, Basse Normandie
  - Clinique St Laurent, Rennes, Basse Normandie
  - Chp St Greg, Saint-Grégoire, Basse Normandie
  - Ch St Malo, St-Malo, Basse Normandie
  - CHG William MOREY, Chalon S/s, Bourgogne-Franche-Comté
  - CHU du BOCAGE, Dijon, Bourgogne-Franche-Comté
  - Clinique St Faron, Meaux, Champagne
  - Cac Jean Godinot, Reims, Champagne
  - Hopital St Quentin, Saint-Quentin, Champagne
  - Hopital Troyes, Troyes, Champagne
  - Clinique Pasteur, Évreux, Haute Normandie
  - CH Jacques Monod, Montivilliers, Haute Normandie
  - CHG, Alès, Languedoc
  - CHG, Carcassonne, Languedoc
  - Chu St Eloi, Montpellier, Languedoc
  - CHU Caremeau, Nîmes, Languedoc
  - Ch Du Pays D'Aix, Aix-en-Provence, Marseille
  - Clinique Rambot, Aix-en-Provence, Marseille
  - Ch Duffaut, Avignon, Marseille
  - Chu Timone, Marseille, Marseille
  - Fondation Saint Joseph, Marseille, Marseille
  - Hopital A.Pare, Marseille, Marseille
  - IPC, Marseille, Marseille
  - Chu Estaing, Clermont, Massif Central
  - Chu Gabriel Montpied, Clermont, Massif Central
  - Pole Sante Republique, Clermont, Massif Central
  - Clinique Vitalia Desertines, Montluçon, Massif Central
  - CHR, Roanne, Massif Central
  - Icl St Etienne, Saint-Etienne, Massif Central
  - CHG Cahors, Cahors, Midi Pyrennees
  - CHG St Gaudens, Saint-Gaudens, Midi Pyrennees
  - Clinique de l'Ormeau, Tarbes, Midi Pyrennees
  - CHU Purpan, Toulouse, Midi Pyrennees
  - Clinique Pasteur, Toulouse, Midi Pyrennees
  - Inst. Claudius Regaud, Toulouse, Midi Pyrennees
  - Clinique des Bonnettes, Arras, Nord
  - CH Boulogne-sur-Mer, Boulogne, Nord
  - Centre Oscar Lambret, Lille, Nord
  - Clinique des Dentellieres, Valenciennes, Nord
  - Chi Frejus - St Raphael, Fréjus, Paca
  - Clinique Belvédère, Nice, Paca
  - CH Sainte Musse, Toulon, Paca
  - H.I.A Saint Anne, Toulon, Paca
  - Victor Dubos, Argenteuil, Paris Nord
  - Clinique Ste Marie, Osny, Paris Nord
  - Saint Antoine, Paris, Paris Nord
  - Saint Louis, Paris, Paris Nord
  - TENON, Paris, Paris Nord
  - Hpt Rene Dubos, Pontoise, Paris Nord
  - BEAUJON, Clichy, Paris Ouest
  - Hopital Mignot, Le Chesnay, Paris Ouest
  - Hopital Franco Britannique, Levallois-Perret, Paris Ouest
  - Hopital Des Courses, Maisons-Laffitte, Paris Ouest
  - HARTMANN, Neuilly/seine, Paris Ouest
  - Hopital Foch, Suresnes, Paris Ouest
  - Ico Angers, Angers, Pays de la Loire Region
  - Ch Le Mans, Le Mans, Pays de la Loire Region
  - Victor Hugo, Le Mans, Pays de la Loire Region